CLINICAL TRIAL: NCT01628913
Title: Randomized Phase II Study of BEZ235 or Everolimus in Advanced Pancreatic Neuroendocrine Tumors
Brief Title: Efficacy and Safety of BEZ235 Compared to Everolimus in Patients With Advanced Pancreatic Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial was terminated based on an interim analysis as BEZ235 did not demonstrate a progression free survival advantage to everolimus treatment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235Z2401; CBEZ235Z2401 (Other: Novartis); 2012-000769-19
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Pancreatic Neuroendocrine Tumors (pNET)
Keywords: Pancreatic; Neuroendocrine tumors; PNET; BEZ235; Everolimus
MeSH Terms: conditions — Neuroendocrine Tumors; Neuroectodermal Tumors, Primitive | interventions — dactolisib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BEZ235 (Experimental): Patients received BEZ235 400 mg bid p.o. (by mouth, twice daily)
  Interventions: Drug: BEZ235
- Everolimus (Active Comparator): Patients received Everolimus 10 mg qd p.o. (by mouth, daily)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: BEZ235 — BEZ235 400 mg bid p.o. (by mouth, twice daily)
  Arms: BEZ235
Drug: Everolimus — Everolimus 10 mg qd p.o. (by mouth, daily)
  Arms: Everolimus

SUMMARY:
This was a multicenter, open label, randomized phase II study to evaluate the efficacy and safety of BEZ235 as compared to everolimus in patients with advanced, low to intermediate grade pancreatic neuroendocrine tumor (pNET).

DETAILED DESCRIPTION:
Patients with advanced (unresectable or metastatic), low to intermediate grade (histologically confirmed well and moderately differentiated) pancreatic neuroendocrine tumor (pNET) were randomized to either BEZ235 or everolimus. The study was planned to include 140 patients, with 70 patients in the BEZ235 treatment group and 70 patients in the everolimus treatment group. An interim analysis was conducted on 62 randomized patients. The study was terminated as the BEZ235 treatment did not demonstrate a progression free survival advantage to everolimus treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced histologically confirmed well differentiated pancreatic neuroendocrine tumor
* Progressive disease within the last 12 months
* Measurable disease per RECIST Version 1.0 determined by multiphase MRI or triphasic CT

Exclusion Criteria:

* Prior treatment with mTOR or PI3K inhibitors
* Patients with more than 2 prior systemic treatment regimens
* Previous cytotoxic chemotherapy, targeted therapy, or biotherapy within the last 4 weeks

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (4):
  - Cedars Sinai Medical Center SC-3, Los Angeles, California
  - University of Colorado Univ Colorado, Aurora, Colorado
  - University of Kentucky Univ Kebtucky, Lexington, Kentucky
  - Montefiore Medical Center SC, The Bronx, New York
- France (5):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
- Italy (3):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
- Novartis Investigative Site, Kazan', Russia
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Lucerne, Switzerland
- United Kingdom (4):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Sheffield

REFERENCES:
- [Derived] Salazar R, Garcia-Carbonero R, Libutti SK, Hendifar AE, Custodio A, Guimbaud R, Lombard-Bohas C, Ricci S, Klumpen HJ, Capdevila J, Reed N, Walenkamp A, Grande E, Safina S, Meyer T, Kong O, Salomon H, Tavorath R, Yao JC. Phase II Study of BEZ235 versus Everolimus in Patients with Mammalian Target of Rapamycin Inhibitor-Naive Advanced Pancreatic Neuroendocrine Tumors. Oncologist. 2018 Jul;23(7):766-e90. doi: 10.1634/theoncologist.2017-0144. Epub 2017 Dec 14. PMID 29242283

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were assigned to one of the following 2 treatment arms in a ratio of 1:1: BEZ235 (investigational arm) or everolimus (control arm)
Period: Overall Study
Arm/Group | BEZ235 | Everolimus
Started | 31 | 31
Completed | 0 | 0
Not Completed | 31 | 31
Not completed — Adverse Event | 12 | 5
Not completed — Disease Progression | 11 | 14
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 1 | 0
Not completed — study terminated by Sponsor | 4 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BEZ235 | Everolimus | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (12.43) [32.0 to 81.0] | 57.8 (11.85) [34.0 to 78.0] | 57.1 (12.07) [32.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until the date of the first radiologically documented disease progression or death due to any cause. PFS is based on local investigator assessment. Patients will be followed up for the duration of the study and for an expected average of every 12 weeks after randomization. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of all target lesions, or unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: up to approx. 18 months
Population: Full analysis set: The Full analysis set (FAS) comprised all patients who were randomized to study treatment. According to the intent to treat principle, patient was analyzed according to the treatment and strata they had been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BEZ235 | Everolimus
Number analyzed (Participants) | 31 | 31
Months | 8.2 [5.3 to NA] — Upper Limit could not be calculated due to insufficient number of events. | 10.8 [8.1 to NA] — Upper Limit could not be calculated due to insufficient number of events.

2. Secondary Outcome: Objective Response Rate
Description: Proportion of patients with a best overall response during the study of complete response (CR) or partial response (PR), based on the investigator assessment. 2. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for all target and non-target lesions, as well as new lesions as assessed by CT or MRI: Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of all target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to approx. 18 months
Population: Trial terminated based on the results of an interim analysis of the primary OM ( which demonstrated BEX235 not having improved PFS (progression free survival) vs everolimus).The secondary OM analyses were not conducted.
Arm/Group | BEZ235 | Everolimus
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to the date of death due to any cause
Time Frame: up to approx. 30 months
Population: as for outcome 2
Arm/Group | BEZ235 | Everolimus
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time from randomization to the date of the first of the following events:death due to any cause or progressive disease, treatment discontinuation due to toxicity or treatment discontinuation due to patient preference
Time Frame: up to approx. 18 months
Population: as for outcome 2
Arm/Group | BEZ235 | Everolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | BEZ235 | Everolimus
Serious Adverse Events (participants affected / at risk) | 11/31 | 9/31
Other Adverse Events (participants affected / at risk) | 31/31 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BEZ235 (N=31) | Everolimus (N=31)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BEZ235 (N=31) | Everolimus (N=31)
Anaemia (Blood and lymphatic system disorders) | 8 | 11
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Palpitations (Cardiac disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 12 | 8
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5
Cheilitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 28 | 17
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 17 | 10
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 0
Proctitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 23 | 20
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 14 | 7
Asthenia (General disorders) | 13 | 13
Face oedema (General disorders) | 0 | 2
Fatigue (General disorders) | 7 | 10
Influenza like illness (General disorders) | 3 | 2
Mucosal inflammation (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 6 | 11
Pyrexia (General disorders) | 9 | 4
Xerosis (General disorders) | 0 | 3
Conjunctivitis (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 5
Oral herpes (Infections and infestations) | 0 | 2
Tooth infection (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 2
Blood cholesterol increased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 6 | 2
Cardiac murmur (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Pancreatic enzymes decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 0 | 7
Weight decreased (Investigations) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 9 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 11
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 6 | 7
Lethargy (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 2 | 1
Depression (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 8
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 11 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Trial terminated based on the results of a pre-planned interim analysis of the primary OM ( which demonstrated BEX235 not having improved PFS (progression free survival) vs everolimus)..The secondary OM analyses were not conducted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.